CLINICAL TRIAL: NCT05503199
Title: Comparison of Strategies for Vascular Access Closure After Transcatheter Aortic Valve Implantation: The ACCESS-TAVI Randomized Trial
Brief Title: Comparison of Strategies for Vascular Access Closure After Transcatheter Aortic Valve Implantation
Acronym: ACCESS-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. T00122
Record Dates: First submitted 2022-08-02; First posted 2022-08-16 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation (TAVI); Vascular Closure Device
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined suture- and plug-based VCD strategy (Experimental): 1 ProGlide or ProStyle + 1 Angio-Seal
  Interventions: Device: Combination of one Perclose ProGlide or ProStyle (Abbott Vascular) and one Angio-Seal (Terumo).
- Pure suture-based VCD strategy (Experimental): 2 ProGlides or ProStyles
  Interventions: Device: Combination of two ProGlides or ProStyles (Abbott Vascular).

INTERVENTIONS:
Device: Combination of one Perclose ProGlide or ProStyle (Abbott Vascular) and one Angio-Seal (Terumo). — Combined suture- and plug-based VCD strategy after TF-TAVI.
  Arms: Combined suture- and plug-based VCD strategy
Device: Combination of two ProGlides or ProStyles (Abbott Vascular). — Pure suture-based VCD strategy after TF-TAVI.
  Arms: Pure suture-based VCD strategy

SUMMARY:
The ACCESS-TAVI trial is an investigator-initiated, prospective, randomized, multicenter, open-label clinical trial. The objective of the trial is to compare two different vascular closure device strategies for large bore vascular access following transfemoral transcatheter aortic valve implantation with regard to safety and efficacy.

DETAILED DESCRIPTION:
Detailed information is provided elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and able to give consent
* Patients with an indication for TF-TAVI as judged by the local multi-disciplinary heart team
* Feasibility of transfemoral access route using commercially available transcatheter heart valves and delivery systems
* Written informed consent

Exclusion Criteria:

* Vascular access site anatomy not suitable for percutaneous vascular closure device
* Vascular access site complications prior to the TAVI procedure
* Known allergy or hypersensitivity to any component of the VCD
* Active bleeding or bleeding diathesis
* Absence of computed tomographic data of the access site before the procedure
* Systemic infection or local infection at or near the access site
* Limited long-term prognosis due to other comorbid conditions
* Patient cannot adhere to or complete the trial protocol for any reason
* Pregnancy
* Participation in any other interventional trial
* Patients with mechanical heart valves in mitral position
* Patients with elevated international normalized ratio (INR) due to oral anticoagulation therapy requiring reversal of vitamin K antagonists prior to TAVI using prothrombin complex concentrate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Major or minor vascular and access-site-related complications or need for additional interventional or surgical procedures related to vascular hemostasis. | In-hospital, in average three days
  The primary outcome measure is a combination of major or minor vascular and access-site-related complications or need for additional interventional (e.g. covered stent implantation) or surgical procedures related to vascular hemostasis according to updated VARC-3 criteria.

SECONDARY OUTCOMES:
Major or minor vascular and access-site-related complications after TF-TAVI. | At 30-day follow-up
  Combination of major or minor vascular and access-site-related complications after TF-TAVI according to VARC-3 criteria.
Individual components of the primary endpoint, namely 1) major or minor vascular and access-site-related complications, 2) need for additional interventional or surgical procedures related to vascular hemostasis. | In-hospital (in average three days) and at 30-day follow-up
  Individual components of the primary endpoint according to VARC-3 criteria.
Unplanned use of endovascular stent and/or vascular surgery or other endovascular interventions at the puncture site. | In-hospital (in average three days) and at 30-day follow-up
  Unplanned use of endovascular stent (e.g. covered stent) and/or vascular surgery or other endovascular interventions at the puncture site.
Any bleedings. | In-hospital (in average three days) and at 30-day follow-up
  Any type of bleedings according to VARC-3 criteria.
Need for blood transfusions. | In-hospital (in average three days)
  Need for blood transfusions for vascular access-site-related bleedings or vascular complications.
Percent diameter stenosis of vascular access vessel. | Intra-procedural
  Percent diameter stenosis of vascular access vessel on post-procedural angiography.
All-cause mortality. | In-hospital (in average three days) and at 30-day follow-up
  All-cause mortality according to VARC-3 criteria.
Length of post-procedural hospital stay. | In-hospital (in average three days)
  Length of post-procedural hospital stay (days).
Time from VCD application to complete hemostasis. | Intra-procedural
  Time from VCD application to complete hemostasis (seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joner, MD, Principal Investigator — Deutsches Herzzentrum München; Tobias Rheude, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No